CLINICAL TRIAL: NCT03207282
Title: Treatment Resistant Depression in America Latina
Acronym: TRAL
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108329; 54135419RSD4001 (Other: Jannsen Cilag S.A.)
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Diagnosis of Depression: Study population consists of participants with a clinical diagnosis of depression, being treated in a psychiatry reference site (example, clinic, ambulatory, hospital, day-hospital) in 4 Latin American countries. Participants with Major Depressive Disorder (MDD) enrolled in Phase 1, will be assessed to estimate the prevalence of Treatment Resistant Depression (TRD) and participants with this diagnosis will be included in Phase 2. Participants with TRD will be followed-up for 1 year.

SUMMARY:
The purpose of this study is to estimate the prevalence of Treatment Resistant Depression (TRD) among Major Depressive Disorder (MDD) participants being treated in a psychiatry reference site (example, clinic, ambulatory, hospital, day-hospital) in 4 Latin American countries: Argentina, Brazil, Colombia and Mexico; and to evaluate all and depression-related healthcare resource utilization in TRD participants.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* Major depressive disorder (MDD) diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV), that was confirmed by MINI International Neuropsychiatric Interview, 5.0 version (MINI)
* Treated or untreated participants with a new or continued episode of depression at the time of the enrolment
* Participants must be capable of completing the corresponding assessments in the study
* Participants must be capable of signing the informed consent form

Phase 2:

* Diagnosis of Treatment Resistant Depression (TRD), to be described by the investigator, based on the criteria:

  1. Adequate follow-up and treatment with at least 2 antidepressants
  2. Without complete response to treatment (based on Montgomery-Asberg Depression Rating Scale [MADRS])

     Exclusion Criteria:
* Participants diagnosed of psychosis, schizophrenia, bipolar disorder, schizoaffective disorder, or dementia
* Participants with substance dependence considered serious by the investigator
* Participant currently participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of participants with Major Depressive Disorder (MDD) being treated in a psychiatry reference site (clinic, ambulatory, hospital, day-hospital) in 4 Latin American countries and will be assessed to estimate the prevalence of Treatment Resistant Depression (TRD) among MDD participants.
Sampling Method: Probability Sample
Enrollment: 1539 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Treatment Resistant Depression (TRD) | Baseline (Day 1)
  Prevalence of TRD will be assessed as percentage of participants with TRD among Major Depressive Disorder (MDD) participants.
Healthcare Resource Utilization in TRD Participants | Up to Month 12
  Healthcare resources utilized in TRD participants will be estimated.

SECONDARY OUTCOMES:
Demographic Characteristics of TRD Participants | Baseline (Day 1)
  Demographic characteristics (such as age and gender) of TRD participants will be assessed at baseline.
Number of Participants With Comorbid Conditions | Baseline (Day 1)
  Comorbid conditions of TRD participants will be assessed at baseline.
Treatment Patterns Over Time for TRD Participants | Baseline (Day 1) up to Month 12
  Treatment patterns of TRD participants will be assessed over time.
Treatment Duration for MDD | Baseline (Day 1) up to Month 12
  Treatment duration is defined as the time interval between baseline and time to next therapy (since the date of the first and second regimen to the start of third regimen).
Treatment Pattern for TRD Participants by Line | Baseline (Day 1) up to Month 12
  Treatment patterns for TRD participants will be determined by distribution of every line of the treatment regimen including pharmaceutical and non-pharmaceutical treatments.
Sequence of Drugs | Baseline (Day 1) up to Month 12
  Sequence of drugs taken by TRD participants will be determined.
Severity of Symptoms as Measured by Montgomery-Asberg Depression Rating Scale (MADRS) Score | Baseline (Day 1), Month 3, 6, 9 and 12
  The MADRS is a 10 item scale for the evaluation of depressive symptoms (Montgomery et al 1979). The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts. Each MADRS item is rated on a 0 to 6 scale with a total score ranging from 0 60. Higher MADRS scores indicate higher levels of depressive symptoms (more severe condition) and lower scores indicate a decreased severity of depression.
Level of Disability as Measured by Sheehan Disability Scale (SDS) | Baseline (Day 1), Month 6, and 12
  SDS is a composite of 3 self-rated items designed to measure the extent to which 3 major sectors in the participant's life are impaired by panic, anxiety, phobic, or depressive symptoms. The participant rates the extent to which his or her (1) work, (2) social life or leisure activities, and (3) home life or family responsibilities are impaired by his or her symptoms on a 10-point visual analog scale. To get a total score add up the 3 individual scores and the total score ranges from "0 = unimpaired" to "30 = highly impaired". Higher scores indicate worsening.
Suicidality Risk (Ideation and Attempts) as Measured by Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Baseline (Day 1), Month 3, 6, 9, and 12
  Suicidal ideation or behavior will be measured using C SSRS score. C-SSRS is a clinician rated assessment of suicidal behavior and/ or intent. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 yes/no items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Worsening of suicidal ideation was an increase in severity of suicidal ideation from baseline.
Healthcare Costs in TRD Participants | Up to Month 12
  Total healthcare costs and healthcare costs related to depression will be determined in TRD participants.
Indirect Cost Associated With Work Productivity Loss | Baseline (Day 1) up to Month 12
  Work productivity loss was measured by Work Productivity and Activity Impairment Questionnaire (WPAI). The WPAI is a validated, self-administered questionnaire that assesses work and activity impairment during the past 7 days. The WPAI produces 4 types of scores: absenteeism (work time missed), presenteeism (impairment at work/reduced on the job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment. The WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Indirect Cost Associated With Daily Functioning Loss | Baseline (Day 1) up to Month 12
  Indirect cost associated with daily functioning loss will be determined.
Indirect Cost Associated With Caregiver Burden | Baseline (Day 1) and Month 12
  Indirect cost associated with caregiver burden will be determined.
Indirect Cost Associated With Quality of Life | Baseline (Day 1) and Month 12
  Quality of life will be measured by EuroQol-5 Dimension (EQ-5D). The EQ-5D descriptive system comprises the following 5 dimensions: Mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 dimensions is divided into 3 levels of perceived problems (Level 1 indicating no problem, Level 2 indicating slight problems, Level 3 indicating extreme problems). The participant selects an answer for each of the 5 dimensions considering the response that best matches his or her health "today." The descriptive system can be represented as a health state. The EQ-VAS self-rating records the respondent's own assessment of his or her overall health status, on a scale of 0 (worst imaginable health state) to 100 (best imaginable health state).

CONTACTS AND LOCATIONS:
Overall Officials: Jannsen Cilag S.A. Clinical Trial, Study Director — Jannsen Cilag S.A.
Locations (33):
- Argentina (5):
  - Fundacion para el Estudio y Tratamiento de las Enfermedades Mentales, Buenos Aires
  - Instituto DAMIC, Córdoba
  - Clinica Privada de Salud Mental Santa Teresa de Ávila, La Plata
  - CESASIN, Mendoza
  - C I A P Centro de investigacion y Asistencia en Psiquiatria, Rosario
- Brazil (10):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Instituto De Neurociencias Dr. Quevedo Hospital Sao Sebastiao, Criciúma
  - Trial Tech Tecnologia em Pesquisas com Medicamentos, Curitiba
  - Universidade Federal Do Ceara, Fortaleza
  - Instituto Bairral de Psiquiatria, Itapira
  - Faculdade de Medicina da Universidade Federal de Pelotas, Pelotas
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Universidade Federal do Rio de Janeiro - Instituto de Psiquiatria, Rio de Janeiro
  - Hospital Universitario Professor Edgar Santos, Salvador
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Colombia (4):
  - HOMO - ESE Hospital Mental de Antioquia, Bello
  - Instituto Colombiano del Sistema Nervioso, Bogotá
  - Centro de Investigaciones del Sistema Nervioso Grupo Cisne Ltda., Bogotá
  - Conciencia S.A.S, Medellín - Antioquia
- Mexico (14):
  - Hospital Psiquiátrico Granja la Salud Tlazolteotl, Ixtapaluca
  - Hospital Aranda de la Parra S A de C V, León
  - Grupo de Estudios Médicos y familiares Carraci SC, Mexico City
  - Estimulación Magnética Transcraneal de México S.C., Mexico City
  - Hospital Psiquiatrico Fray Bernardino Alvarez, Mexico City
  - Instituto Nacional de Psiquiatria Ramon de la Fuente Muniz, Mexico City
  - Clínica de Neuropsiquiatría Tlatelolco ISSSTE, Mexico City
  - Instituto Nacional de Neurología y Neurocirugía, México
  - Privarte Practice of Dr. Javier Zambrano, México
  - Instituto Jalisciense de Salud Mental, México
  - Centro para las Adicciones y Salud Mental S.A. de C.V., Monterrey
  - cit NEUROPSIQUE, Monterrey
  - Hospital Central Dr Ignacio Morones Prieto, San Luis Potosí City
  - Clínica de Consulta Externa Alfredo del Mazo Vélez ISSEMyM, Toluca

REFERENCES:
- [Derived] Soares B, Kanevsky G, Teng CT, Perez-Esparza R, Bonetto GG, Lacerda ALT, Uribe ES, Cordoba R, Lupo C, Samora AM, Cabrera P. Prevalence and Impact of Treatment-Resistant Depression in Latin America: a Prospective, Observational Study. Psychiatr Q. 2021 Dec;92(4):1797-1815. doi: 10.1007/s11126-021-09930-x. Epub 2021 Aug 31. PMID 34463905